CLINICAL TRIAL: NCT05163405
Title: Perspectives of Subcutaneous Velcade at Home of Patients With Myeloma.
Status: Completed | Type: Observational
Sponsor: Karin B. Ø. Dieperink (Other)
Responsible Party: Sponsor-Investigator, Karin B. Ø. Dieperink, Nurse, PhD, Associate Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: Velcade at home
Record Dates: First submitted 2021-12-03; First posted 2021-12-20 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Bortezomib — Self-administration of subcutaneously Velcade.
  Other Names: Velcade

SUMMARY:
In the present study, we have trained 10 patients in subcutaneous self-administration of Velcade. After their training, patients will alternately receive their treatment in the hospital and at home by self-administration. In keeping with common practice, a nurse contacts the patients by telephone before 9.00 am on the day of treatment to ensure that the patient is physically "fit" to receive the medication and to discuss any side effects. To highlight the advantages and disadvantages of the changed treatment practice from the perspectives of both patients and healthcare professionals, data is collected from two consecutive semi-structured interviews with n = 10 patients and n = 1 focus group interview of the healthcare professionals involved. Moreover, time registration of medication administration both at the hospital and in the patients' home is done. The qualitative data will be analyzed via the method of condensation and continual quantitative data will form the basis of a cost-benefit analysis.

ELIGIBILITY:
Inclusion criteria

* Patients must have Multiple Myeloma
* Patients (or their relatives) must be deemed physically and cognitively suitable and willing for self-administration of subcutaneous Velcade
* Patients must be able to understand and speak Danish
* Patients must have received a minimum of 1 treatment cycle in the outpatient clinic

Exclusion criteria

* Lack of willingness to participate in scheduled interviews
* Patients who are cognitively affected
* Must not be receiving trial treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Multiple Myeloma in treatment with Velcade in Department of Hematology X, outpatient clinic, at Odense University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Patients experience of self-administration of Velcade | Through study completion, from 01. dec. 2019 until 01. jun. 2022
  Qualitative interviews with all 10 included patients

SECONDARY OUTCOMES:
Organizational perspective | Through study completion, from 01. dec. 2019 until 01. jun. 2022
  Patients and health professionals (including pharmacy staff) registration of time spend on treatment on all 10 included patients.
Health care perspective | Through study completion, from 01. dec. 2019 until 01. jun. 2022
  Focus group interview with healthcare professionals involved in the treatment.
Financial perspective | Through study completion, from 01. dec. 2019 until 01. jun. 2022
  Evaluation of financial savings on home treatment including healthcare salaries and transportation.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Brochstedt Dieperink, RN, Study Director — Odense University Hospital. Department of Oncology.
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No